CLINICAL TRIAL: NCT00342797
Title: Retinoblastoma Biomarker Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999993033; OH93-NC-N033
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Retinoblastoma; Melanoma; Sarcoma
Keywords: second primary cancer; retinoblastoma; RB1 germline mutation; Natural History
MeSH Terms: conditions — Retinoblastoma; Melanoma; Sarcoma; Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retinoblastoma cohort: Retinoblastoma patients treated at two hospitals in New York and one hospital in Boston from 1914-2006.

SUMMARY:
Retinoblastoma is a rare pediatric ocular tumor caused by germline and/or somatic mutations in the tumor suppressor gene RB1. Survivors of retinoblastoma, particularly those with the hereditary form of the disease (germline RB1 mutations) are highly susceptible to developing additional malignancies, which are a major cause of morbidity and mortality. Since 1984, REB has followed a cohort of 2136 (including 1,995 one-year) retinoblastoma survivors to investigate the contributions of treatment and genetic risk factors to second cancer etiology. The last systematic follow-up for second cancer incidence and cause-specific mortality was completed in 2009. As the cohort ages, we now propose to conduct another interview survey to collect information on newly diagnosed second cancers. Additionally, we propose to expand collection of germline DNA for additional molecular studies in survivors. Retinoblastoma survivors have now entered adult ages when epithelial tumors would be expected to occur with greater frequency. Given that the somatic mutations in the RB1 pathway have been identified in several epithelial tumors (bladder, brain, breast, esophagus, liver, lung, prostate) in addition to sarcomas, it is important to collect new information on these epithelial tumors, and to investigate whether the previously identified high risks of sarcomas and melanoma will persist as the cohort ages. Additionally, our understanding of genetic susceptibility to second cancers is limited. Given that this is the only cohort of long-term survivors of retinoblastoma being followed in the U.S., combined with the leadership role of REB in the study of second cancers, continued follow-up of this cohort will provide unique clinical and epidemiologic data on the long-term cumulative risk of second cancers in this distinctive cohort of childhood cancer survivors.

DETAILED DESCRIPTION:
Retinoblastoma is a rare pediatric ocular tumor caused by germline and/or somatic mutations in the tumor suppressor gene RB1. Survivors of retinoblastoma, particularly those with the hereditary form of the disease (germline RB1 mutations) are highly susceptible to developing additional malignancies, which are a major cause of morbidity and mortality. Since 1984, REB has followed a cohort of 2136 (including 1,995 one-year) retinoblastoma survivors to investigate the contributions of treatment and genetic risk factors to second cancer etiology. The last systematic follow-up for second cancer incidence and cause-specific mortality was completed in 2009. As the cohort ages, we now propose to conduct another interview survey to collect information on newly diagnosed second cancers. Additionally, we propose to expand collection of germline DNA for additional molecular studies in survivors. Retinoblastoma survivors have now entered adult ages when epithelial tumors would be expected to occur with greater frequency. Given that the somatic mutations in the RB1 pathway have been identified in several epithelial tumors (bladder, brain, breast, esophagus, liver, lung, prostate) in addition to sarcomas, it is important to collect new information on these epithelial tumors, and to investigate whether the previously identified high risks of sarcomas and melanoma will persist as the cohort ages. Additionally, our understanding of genetic susceptibility to second cancers is limited. Given that this is the only cohort of long-term survivors of retinoblastoma being followed in the U.S., combined with the leadership role of REB in the study of second cancers, continued follow-up of this cohort will provide unique clinical and epidemiologic data on the long-term cumulative risk of second cancers in this distinctive cohort of childhood cancer survivors.

ELIGIBILITY:
* INCLUSION CRITERIA:

Children treated for retroblastoma over the past 30-plus years.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Survivors of retinoblastoma treated at hospitals in New York City and Boston between 1914-2006 and US residents.
Sampling Method: Non-Probability Sample
Enrollment: 2136 (Actual)
Dates: Start 1993-11-17; Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Mutation in RB1 gene | once
  Location of mutation in the RB1 gene
Subsequent Cancer | At least one year after retinoblastoma
  Risk of subsequent cancer in relation to prior treatment and RB1 mutation

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay M Morton, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (4):
- United States (4):
  - National Cancer Institute (NCI), Bethesda, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Social Scientific Systems, Inc., Durham, North Carolina

REFERENCES:
- [Background] Wong JR, Morton LM, Tucker MA, Abramson DH, Seddon JM, Sampson JN, Kleinerman RA. Risk of subsequent malignant neoplasms in long-term hereditary retinoblastoma survivors after chemotherapy and radiotherapy. J Clin Oncol. 2014 Oct 10;32(29):3284-90. doi: 10.1200/JCO.2013.54.7844. Epub 2014 Sep 2. PMID 25185089
- [Background] Kleinerman RA, Tucker MA, Sigel BS, Abramson DH, Seddon JM, Morton LM. Patterns of Cause-Specific Mortality Among 2053 Survivors of Retinoblastoma, 1914-2016. J Natl Cancer Inst. 2019 Sep 1;111(9):961-969. doi: 10.1093/jnci/djy227. PMID 30698734
- [Background] Kleinerman RA, Schonfeld SJ, Sigel BS, Wong-Siegel JR, Gilbert ES, Abramson DH, Seddon JM, Tucker MA, Morton LM. Bone and Soft-Tissue Sarcoma Risk in Long-Term Survivors of Hereditary Retinoblastoma Treated With Radiation. J Clin Oncol. 2019 Dec 10;37(35):3436-3445. doi: 10.1200/JCO.19.01096. Epub 2019 Oct 17. PMID 31622129